CLINICAL TRIAL: NCT02969265
Title: A Phase-3 Randomized, Double-Blind, Parallel-Group Efficacy and Safety Study Evaluating the Fixed-Dose Combination of Candesartan Plus Amlodipine (8/5 mg) in Chinese Subjects With Mild/Moderate Essential Hypertension, Who Do Not Achieve Target Blood Pressure Following Treatment With Amlodipine 5 mg Monotherapy
Brief Title: An Efficacy and Safety Study Evaluating the Fixed-Dose Combination of Candesartan Plus Amlodipine in Participants With Mild/Moderate Essential Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons unrelated to product safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCV-116CCB_302; U1111-1184-7520 (Registry Identifier: WHO); CTR20160750 (Registry Identifier: CFDA)
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Hypertension
Keywords: Drug therapy
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCV-116CCB (Candesartan 8 mg Plus Amlodipine 5 mg) (Experimental): Run-in Period: TCV-116CCB placebo-matching tablets, orally, once daily along with amlodipine placebo-matching capsules, orally, once daily up to 2 weeks.
  Single-blind monotherapy treatment period: TCV-116CCB placebo-matching tablets, orally, once daily along with amlodipine 5 mg capsules, orally, once daily up to 4 weeks.
  Double-blind treatment period: TCV-116CCB 8/5 mg tablets, orally, once daily along with amlodipine placebo-matching capsules, orally, once daily up to 8 weeks.
  Interventions: Drug: Amlodipine; Drug: TCV-116CCB; Drug: Amlodipine Placebo; Drug: TCV-116CCB Placebo
- Amlodipine 5 mg (Experimental): Run-in Period: TCV-116CCB placebo-matching tablets, orally, once daily along with amlodipine placebo-matching capsules, orally, once daily up to 2 weeks.
  Monotherapy treatment period: TCV-116CCB placebo-matching tablets, orally, once daily along with amlodipine 5 mg capsules, orally, once daily up to 4 weeks.
  Double-blind treatment period: Amlodipine 5 mg capsules, orally, once daily along with TCV-116CCB placebo-matching tablets, orally, once daily up to 8 weeks.
  Interventions: Drug: Amlodipine; Drug: Amlodipine Placebo; Drug: TCV-116CCB Placebo

INTERVENTIONS:
Drug: Amlodipine — Amlodipine Capsules
Drug: TCV-116CCB — TCV-116CCB Tablets
  Arms: TCV-116CCB (Candesartan 8 mg Plus Amlodipine 5 mg)
Drug: Amlodipine Placebo — Amlodipine placebo-matching capsules
Drug: TCV-116CCB Placebo — TCV-116CCB 8/5 mg placebo-matching tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TCV-116CCB (candesartan cilexetil and amlodipine besylate fixed-dose combination) in Chinese participants with mild to moderate hypertension who do not reach target blood pressure following 4 weeks of treatment with amlodipine monotherapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called TCV-116CCB (candesartan cilexetil and amlodipine besylate fixed-dose combination). This study will look at blood pressure in Chinese participants with grade 1 or 2 essential hypertension.

The study will enroll approximately 370 patients. Prior to the start of study treatment, participants will undergo run-in period of 2 weeks followed by single-blind treatment period of 4 weeks. Upon completion of single-blind treatment period, participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Amlodipine 5 mg
* TCV-116CCB (Candesartan 8 mg Plus Amlodipine 5 mg)

All participants will be asked to take one tablet/capsule at the same time each day throughout the study up to 8 weeks.

This multicenter trial will be conducted China. The overall time to participate in this study is 19 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone plus a final visit 14 days after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has grade 1 or 2 essential hypertension which is not adequately controlled, as defined by mean, trough, sitting, clinic systolic blood pressure (SBP):

   1. ≥155 to <180 mm Hg in participants who have not received any antihypertensive medication in the 14 days prior to Visit 1.
   2. ≥145 to ≤170 mm Hg in participants taking 1 antihypertensive medication at Visit 1.
   3. ≥140 to <160 mm Hg in participants taking 2 antihypertensive medications at Visit 1.
2. Is willing to discontinue current antihypertensive medications.

   Entering amlodipine 5 mg monotherapy:
3. Must have a clinic SBP measurement of 155 to 179 mm Hg inclusive (determined by the mean of 3 sitting, trough, measurements on Day -28, using same arm throughout study) to qualify for entry in to the 4 week single-blind amlodipine 5 mg monotherapy treatment period.

   At double-blind randomization:
4. Has not achieved target blood pressure (defined as clinic SBP ≥140 mm Hg as determined by the mean of 3 sitting, trough, measurements) following 4 weeks single-blind treatment with amlodipine 5 mg monotherapy at Day 1 prior to randomization to double-blind treatment.

Exclusion Criteria:

1. Has clinic SBP ≥180 mm Hg or DBP ≥110 mm Hg.
2. The participant's 3 SBP measurements differ by more than 15 mm Hg (confirmed by a second set of three measurements).
3. Has been randomized/enrolled in an amlodipine or candesartan or candesartan/amlodipine Fixed dose combination study.
4. Has secondary hypertension of any etiology (e.g., renovascular disease documented as the cause of hypertension, pheochromocytoma, Cushing's syndrome).
5. Has any history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, persistent or permanent atrial fibrillation or transient ischemic attack.
6. Has clinically significant cardiac conduction defects (e.g., third-degree atrioventricular block, sick sinus syndrome).
7. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease or hypertrophic cardiomyopathy.
8. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of single-blind amlodipine monotherapy study drug. (This criterion does not apply to those participants with basal cell or Stage 1 squamous cell carcinoma of the skin).
9. Has poorly-controlled type 1 or 2 diabetes mellitus (hemoglobin A1c [HbA1c] >8.0%) at Screening.
10. Has severe renal dysfunction or disease (based on estimated Glomerular filtration rate [GFR] <30 mL/min/1.73m^2) at Screening.
11. Has hypokalemia or hyperkalemia (defined as serum potassium outside of the normal reference range) at Screening.
12. Has an alanine aminotransferase or aspartate aminotransferase level >2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
13. Works a night (third) shift (defined as 10 PM [2200] to 6 AM [0600]) (Only for participants with ambulatory blood pressure monitoring [ABPM]).
14. Has an upper arm circumference <24 cm or >42 cm (Only for participants with ABPM).

    Entering amlodipine 5 mg monotherapy period:
15. Has a clinic SBP ≥180 mm Hg or DBP ≥110 mm Hg.
16. Is non-compliant (<80% or >120%) with study medication during the placebo run-in period.

    Post-single-blind amlodipine 5 mg treatment period:
17. Achieves target blood pressure (defined as clinic SBP<140 mm Hg as determined by the mean of 3 sitting, trough measurements) following 4 weeks single-blind treatment with amlodipine 5 mg monotherapy at Day 1, prior to randomization to double-blind treatment.
18. Has a clinic SBP ≥180 mm Hg or/and DBP ≥110 mm Hg.
19. Is non-compliant (<80% or >120%) with study medication during the amlodipine 5 mg single-blind treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-09 (Estimated); Primary Completion 2018-07-12 (Estimated); Study Completion 2018-07-26 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Trough, Sitting, Clinic Systolic Blood Pressure (SBP) at Week 8 | Baseline and Week 8
  The change between trough SBP measured at Week 8 relative to baseline. It is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.

SECONDARY OUTCOMES:
Change From Baseline in Trough, Sitting, Clinic Diastolic Blood Pressure (DBP) at Week 8 | Baseline and Week 8
  The change between trough DBP measured at Week 8 relative to baseline. It is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Percentage of Participants who Achieved Target Blood Pressure at Week 8 | Week 8
  Target blood pressure is defined as trough, sitting clinic SBP <140 mm Hg, trough, sitting, clinic DBP <90 mm Hg or achieving both trough, sitting clinic SBP (<140 mm Hg) and DBP targets (<90 mm Hg).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (25):
- China (25):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing first hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - The Xiangya Hospitalof Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jilin Siping Central Hospital, Siping, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - the Central Hospital of Xuhui District, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Putuo Center Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan Univeisity, Chengdu, Sichuan
  - Sir Run Run Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Lishui Hospital of Zhejiang Province, Lishui, Zhejiang